CLINICAL TRIAL: NCT01220661
Title: Phase 2 Study of One Dose Prophylactic Antibiotic in Laparoscopic Colorectal Surgery
Brief Title: Safety and Efficacy of One Dose Prophylactic Antibiotic in Laparoscopic Colorectal Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Ji Won Park, M.D., National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-10-485
Record Dates: First submitted 2010-10-12; First posted 2010-10-14 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Colorectal Surgery
Keywords: Colorectal Surgery; Surgical Wound Infection; Laparoscopy; Anti-Bacterial Agents
MeSH Terms: conditions — Surgical Wound Infection | interventions — Cefotetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- One dose (Experimental): One dose prophylactic antibiotic
  Interventions: Drug: Cefotetan

INTERVENTIONS:
Drug: Cefotetan — preoperative one dose prophylactic antibiotic (2g iv, within 1 hour before skin incision)
  Other Names: Yamatetan

SUMMARY:
In colorectal surgery, the use of prophylactic antibiotics is recommended. The standard use of antibiotics for colorectal surgery is three doses.

It has been reported that the surgical site infection rates of laparoscopic colorectal surgery are lower than open colorectal surgery. However, the evidence of proper application of antibiotic for laparoscopic colorectal surgery is still not enough.

The investigators are researching the efficacy and safety of one dose prophylactic antibiotic in laparoscopic colorectal surgery.

DETAILED DESCRIPTION:
In colorectal surgery, the use of prophylactic antibiotics is recommended. The standard use of antibiotics for colorectal surgery is three doses.

One randomized controlled study reported that surgical site infection rates of three doses prophylactic antibiotics are lower than those of one dose in colorectal surgery (4.3 versus 14.2%). But, surgical site infection rates between one dose and three doses were not different in laparoscopic subgroup of this study (11 versus 11%)

It has been reported that the surgical site infection rates of laparoscopic colorectal surgery are lower than open colorectal surgery. However, the evidence of proper application of antibiotic for laparoscopic colorectal surgery is still not enough.

The investigators are researching the efficacy and safety of one dose prophylactic antibiotic in laparoscopic colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients have laparoscopic colorectal surgery for cancer at National Cancer Center
* Patients should sign a written informed consent
* Age between 18-80 years
* Adequate bone marrow function Hb ≥ 10g/dl (after treatment for simple iron deficiency anemia) WBC ≥ 3,000/mm3 PLT ≥ 100,000/mm3
* Adequate kidney function Creatinine ≤ 1.5 mg/dl
* No remarkable evidence of heart dysfunction and lung dysfunction

Exclusion Criteria:

* Patients undergo emergency surgery with multiple symptoms
* Open colorectal surgery for cancer or conversion to an open procedure
* Patients who undergo only ostomy surgery
* Palliative surgery
* Surgery combined with other organs
* Patients on treatment with recurred cancer
* Patients who have active bacterial infection and required parenteral antibiotics
* Patients have an allergy to Cefoxitin
* Other organ cancer history(except who had radical excision for skin cancer)
* Presence of other serious disease
* Mentally ill patients
* Legally unable to participate in clinical trial
* Lactating or pregnant women
* Patients who will obviously fail to regular follow-up visit or will be off study voluntarily
* Not eligible to participate for other reasons by doctor's decision

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2010-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Surgical site infection | Three weeks after surgery
  any surgical infections (superficial incisional infection or infection of deep incision space or organ space infection)

SECONDARY OUTCOMES:
Overall infection | Three weeks after surgery
  Overall infection including surgical site infection, pneumonia, urinary tract infection etc.

CONTACTS AND LOCATIONS:
Overall Officials: Jae Hwan Oh, Principal Investigator — Center for Colorectal Cancer, National Cancer Center Korea
Locations (1):
- National Cancer Center Hospital, Goyang-si, Gyeonggi-do, South Korea